CLINICAL TRIAL: NCT02756897
Title: A Phase II Study of Venetoclax and Ibrutinib in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Venetoclax and Ibrutinib in Treating Patients With Chronic or Small Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0860; NCI-2016-00797 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0860 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, venetoclax) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Beginning on day 1 of cycle 4, patients also receive venetoclax PO QD on days 1-28. Treatment repeats every 28 days for up to 27 cycles in the absence of disease progression or unacceptable toxicity. Patients with residual disease or who are positive for MRD after cycle 27 may continue treatment with ibrutinib.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well venetoclax and ibrutinib work in treating patients with chronic or small lymphocytic leukemia. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving venetoclax and ibrutinib may help control chronic or small lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Estimate therapeutic activity (best response [complete response (CR)/complete response with incomplete recovery (CRi)]) of combined ibrutinib and venetoclax in patients with chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL).

SECONDARY OBJECTIVES:

I. To determine the safety of this combination strategy. II. To estimate the time to best response with this combination. III. To determine the progression-free survival (PFS) and overall survival (OS).

IV. To test pharmacodynamic endpoints and molecular interactions between these two drugs.

V. To assess the therapeutic activity (best response [CR/CRi]) in subgroups of patients defined by immunoglobulin heavy chain variable (IGHV) mutation or fluorescence in situ hybridization (FISH) subtype.

EXPLORATORY OBJECTIVE:

I. To study immunological and molecular changes in the peripheral blood and the bone marrow in response to ibrutinib and venetoclax.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Beginning on day 1 of cycle 4, patients also receive venetoclax PO QD on days 1-28. Treatment repeats every 28 days for up to 27 cycles in the absence of disease progression or unacceptable toxicity. Patients with residual disease or who are positive for minimal residual disease (MRD) after cycle 27 may continue treatment with ibrutinib.

After completion of study treatment, patients are followed up every 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of CLL/SLL:

  * Cohort 1: Refractory to and/or relapsed after at least one prior therapy will be eligible
  * Cohort 2: Untreated patients with high-risk features (del(17p), or mutated TP53, or del(11q), or unmutated IGHV, or >= 65 years of age) are eligible (cohort 2) provided they have active disease requiring treatment as defined by the International Working Group for CLL (IWCLL)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or =< 3 x ULN for patients with Gilbert's disease (in patients [pts] with elevated total bilirubin due to increased indirect bilirubin, pts with direct bilirubin =< 1.5 x ULN are eligible)
* Creatinine clearance > 50 mL/min (calculated according to institutional standards or using Cockcroft-Gault, Modification of Diet in Renal Disease [MDRD], or Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x ULN, unless clearly due to disease involvement
* Platelet count of greater than 20,000/mul, with no platelet transfusion in 2 weeks prior to registration; this criteria is waived if the thrombocytopenia is due to bone marrow involvement with the disease
* Women of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (beta-hCG) pregnancy test result within 7 days prior to the first dose of study drugs and must agree to use an effective contraception method during the study and for 30 days following the last dose of study drug; women of non- childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy; men who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
* Free of prior malignancies for 2 years with exception of patients diagnosed with basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast, who are eligible even if they are currently treated or have been treated and/or diagnosed in the past 2 years prior to study enrolment; if patients have another malignancy that was treated within the last 2 years, such patients may be enrolled if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center, and after consultation with the principal investigator
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* Major surgery, radiotherapy, chemotherapy, biologic therapy, immunotherapy, investigational therapy within 3 weeks prior to the first dose of the study drugs
* Uncontrolled active systemic infection (viral, bacterial, and fungal)
* Known positive serology for human immunodeficiency virus (HIV), due to potential drug-drug interactions between anti-retroviral medications and the study drugs
* Active hepatitis B infection (defined as the presence of detectable hepatitis B virus [HBV] deoxyribonucleic acid [DNA], hepatitis B e [HBe] antigen or hepatitis B surface [HBs] antigen); subjects with serologic evidence of prior vaccination (hepatitis B surface antigen [HBsAg] negative, anti-HBs antibody positive, anti-hepatitis B core [HBc] antibody negative) are eligible; patients who are HBsAg negative/hepatitis B surface antibody (HBsAb) positive but hepatitis B core antibody (HBcAb) positive are eligible, provided HBV DNA is negative
* Active hepatitis C, defined by the detectable hepatitis C ribonucleic acid (RNA) in plasma by polymerase chain reaction (PCR)
* Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune thrombocytopenia) requiring steroid therapy with > 20 mg daily of prednisone dose or equivalent
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 2 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Patient is pregnant or breast-feeding
* Concurrent use of warfarin
* Received strong (CYP3A) inhibitors or strong CYP3A inducers within 7 days of starting study drugs
* Consumed grapefruit, grapefruit products, Seville oranges, or star fruit within 7 days of starting study drugs
* Prior treatment with venetoclax or ibrutinib
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Best response (complete response /complete response with incomplete recovery) of combined ibrutinib and venetoclax | Up to 2 months after treatment
  For each cohort, the best response (complete response /complete response with incomplete recovery) rate will be estimated along with the exact 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of toxicities | Up to 6 weeks of treatment
  Will be defined as prolonged neutropenia or thrombocytopenia lasting > 42 days; febrile neutropenia; hospitalization due to infection; early death; major bleeding due to thrombocytopenia. Will be monitored in each disease cohort separately using the Bayesian method of Thall, Simon and Estey. Safety data will be summarized using descriptive statistics.
Time to response with combination of ibrutinib and venetoclax | Up to 8 years
  Estimated using the Kaplan-Meier method in each cohort.
Overall survival | Up to 8 years
  Estimated using the Kaplan-Meier method in each cohort.
Progression-free survival | Up to 8 years
  Estimated using the Kaplan-Meier method in each cohort.
Complete response/complete response with incomplete recovery rate in each subgroups of patients | Up to 8 years
  Will be defined by IGHV mutation or fluorescence in situ hybridization (FISH) subtype. Will be estimated along with the exact 95% confidence interval.

OTHER OUTCOMES:
Changes in immunological biomarkers | Up to 8 years
  Will be summarized over time and will be assessed using linear or non-linear mixed effect models as appropriate.
Changes in molecular biomarkers | Up to 8 years
  Will be summarized over time and will be assessed using linear or non-linear mixed effect models as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain N, Keating M, Thompson P, Ferrajoli A, Burger JA, Borthakur G, Takahashi K, Estrov Z, Sasaki K, Fowler N, Kadia T, Konopleva M, Alvarado Y, Yilmaz M, DiNardo C, Bose P, Ohanian M, Pemmaraju N, Jabbour E, Kanagal-Shamanna R, Patel K, Wang W, Jorgensen J, Wang SA, Garg N, Wang X, Wei C, Cruz N, Ayala A, Plunkett W, Kantarjian H, Gandhi V, Wierda WG. Ibrutinib Plus Venetoclax for First-line Treatment of Chronic Lymphocytic Leukemia: A Nonrandomized Phase 2 Trial. JAMA Oncol. 2021 Aug 1;7(8):1213-1219. doi: 10.1001/jamaoncol.2021.1649. PMID 34110383
- [Derived] Jain N, Keating M, Thompson P, Ferrajoli A, Burger J, Borthakur G, Takahashi K, Estrov Z, Fowler N, Kadia T, Konopleva M, Alvarado Y, Yilmaz M, DiNardo C, Bose P, Ohanian M, Pemmaraju N, Jabbour E, Sasaki K, Kanagal-Shamanna R, Patel K, Jorgensen J, Garg N, Wang X, Sondermann K, Cruz N, Wei C, Ayala A, Plunkett W, Kantarjian H, Gandhi V, Wierda W. Ibrutinib and Venetoclax for First-Line Treatment of CLL. N Engl J Med. 2019 May 30;380(22):2095-2103. doi: 10.1056/NEJMoa1900574. PMID 31141631
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org